CLINICAL TRIAL: NCT00005915
Title: A Randomized Study of a Prescribed 4-Month Structured Treatment Interruption (STI) Followed by Initiation of a New Antiretroviral Regimen Versus Immediate Initiation of a New Antiretroviral Regimen in HIV-Infected Patients With Multidrug Resistant (MDR) Virus
Brief Title: A Comparison of Two Anti-HIV Treatment Plans
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 064; 11619 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2000-06-15; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Administration Schedule; Drug Resistance, Microbial; Disease Progression; Genotype; Phenotype; Drug Resistance, Multiple; Anti-HIV Agents; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Disease Progression

SUMMARY:
The purpose of this study is to compare 2 treatment plans to try to increase the effects of anti-HIV drugs in patients who are resistant to the drug effects.

Sometimes the increase in a patient's viral load (the level of HIV in the blood) can be slowed or stopped by taking anti-HIV drugs. This does not always happen. Sometimes anti-HIV drugs work at first but then stop working. When most of the usual anti-HIV drugs no longer seem to work, the virus is called multidrug-resistant (MDR). This study will compare 2 treatment plans to try to increase the effects of anti-HIV drugs in patients with MDR virus.

DETAILED DESCRIPTION:
An increasing number of patients are developing multidrug-resistant (MDR) virus, as determined by genotypic antiretroviral resistance testing (GART), due to treatment failure to suppress viral replication after several rounds of combination antiretroviral therapy. The best therapeutic strategy for these patients is uncertain. Two strategies currently being used are (1) STI followed by a new antiretroviral regimen and (2) immediate initiation of a new antiretroviral regimen.

Patients are screened for the presence of MDR virus and a plasma HIV RNA level greater than 10,000 [AS PER AMENDMENT 07/03/01: greater than 5,000] copies/ml. Eligible patients attend a baseline visit [AS PER AMENDMENT 07/03/01: and a subsequent randomization visit] where the qualifying GART results are provided. Patients who consent to participate have phenotypic antiretroviral resistance testing (PART) done on a specimen from the same blood draw that was used for the GART evaluation. After PART results are available, patients are randomized [AS PER AMENDMENT 07/03/01: If the predicted sensitivities are not available for some or all drugs included in the PART, the patient may still be randomized.] to either a 4-month STI followed by a new antiretroviral regimen or an immediate new antiretroviral regimen. The antiretroviral regimens chosen are based on the patients' history and both GART and PART results. [AS PER AMENDMENT 07/03/01: Additional GART and PART may be requested after at least 4 months of antiretroviral treatment.] Patients have the follow-up data collection done at Months 1-8 and every 4 months thereafter. Changes in antiretroviral therapy, Grade 4 adverse experiences, progression of disease, and deaths are reported as they occur. Patients are seen for clinical management as often as deemed necessary. All patients are followed to a common closing date estimated to be 24 months after the last patient is randomized. Some patients may participate in a Point Mutation Substudy [AS PER AMENDMENT 07/03/01: Plasma Point Mutation Substudy and PBMC Point Mutation Substudy].

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible if they:

* Have proof of MDR virus from a blood test.
* Have a viral load above 5,000 copies/ml from the same blood sample showing MDR virus.
* Intend to start a new anti-HIV treatment around the time of the study.
* Have been on a stable anti-HIV treatment between 14 days prior to the blood test mentioned above and when they are randomly assigned to a treatment.
* Are at least 13 years old (consent of parent or guardian required if under 18).
* (This protocol has been changed to reflect new criteria.)

Exclusion Criteria

Patients will not be eligible if they:

* Have received a vaccine or had an illness that might affect viral load within 14 days before the blood test showing MDR virus.
* Have received IL-2 within 4 months of the above-mentioned blood test or plan to take IL-2 during the study.
* Have an opportunistic (AIDS-related) infection requiring treatment.
* Are pregnant or breast-feeding.
* Are currently participating in CPCRA 057 (PIP study).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480
Dates: Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jody Lawrence, Study Chair
Locations (21):
- United States (21):
  - Community Consortium / UCSF, San Francisco, California
  - Lawrence Goldyn, MD, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Univ Hosp Infectious Disease, Denver, Colorado
  - Yale U / New Haven Med Ctr / AIDS Clinical Trials Unit, New Haven, Connecticut
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Our Lady of the Lake Regional Med Ctr, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Clinical Trials, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - Bronx-Lebanon Hosp Ctr, The Bronx, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Montrose Clinic, Houston, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Univ TX Health Science Ctr, Houston, Texas
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Background] Lawrence J, Mayers DL, Hullsiek KH, Collins G, Abrams DI, Reisler RB, Crane LR, Schmetter BS, Dionne TJ, Saldanha JM, Jones MC, Baxter JD; 064 Study Team of the Terry Beirn Community Programs for Clinical Research on AIDS. Structured treatment interruption in patients with multidrug-resistant human immunodeficiency virus. N Engl J Med. 2003 Aug 28;349(9):837-46. doi: 10.1056/NEJMoa035103. PMID 12944569
- [Result] Anti-HIV agents. An attempt at treatment interruption--trial CPCRA 064. TreatmentUpdate. 2003 Aug-Sep;15(5):4-5. No abstract available. PMID 17216857
- [Result] Lawrence J, Hullsiek KH, Thackeray LM, Abrams DI, Crane LR, Mayers DL, Jones MC, Saldanha JM, Schmetter BS, Baxter JD. Disadvantages of structured treatment interruption persist in patients with multidrug-resistant HIV-1: final results of the CPCRA 064 study. J Acquir Immune Defic Syndr. 2006 Oct 1;43(2):169-78. doi: 10.1097/01.qai.0000242450.74779.ee. PMID 16951642
- [Result] Paquet AC, Baxter J, Weidler J, Lie Y, Lawrence J, Kim R, Bates M, Coakley E, Chappey C. Differences in reversion of resistance mutations to wild-type under structured treatment interruption and related increase in replication capacity. PLoS One. 2011 Jan 31;6(1):e14638. doi: 10.1371/journal.pone.0014638. PMID 21297946